CLINICAL TRIAL: NCT06125249
Title: Humanin's Value for Early Diagnosis and Short-term Prognosis in Patients With AKI After Heart Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Li zhilian (Other)
Responsible Party: Sponsor-Investigator, Li zhilian, Deputy Chief Physician, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Other Study IDs: KJ012019455
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Acute Kidney Injury; Heart Transplant Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with AKI after heart transplantation: AKI occurs in patients after heart transplantation
- Patients did not develop AKI after heart transplantation: Patients who do not develop AKI after heart transplantation

SUMMARY:
The goal of this observational study is to explore the value of Humanin for early diagnosis and short-term prognosis of AKI patients after heart transplantation. The main question it aims to answer are:whether Humanin can be a novel marker for predicting AKI after heart transplantation Researchers will compare the Humanin concentration in patients with AKI did not occur after heart transplantation to see if Humanin can be a novel marker for predicting AKI after heart transplantation

DETAILED DESCRIPTION:
Heart transplantation is an important means of treating end-stage heart disease, acute kidney injury is a common complication after heart transplantation, can lead to perioperative and early postoperative patient death, can also lead to the development of chronic kidney disease after heart transplantation, and even progress to ESRD, the literature reports that the incidence of acute kidney injury after heart transplantation is 14% ~ 76%, resulting in severe renal impairment and the proportion requiring dialysis treatment is 5% ~ 39%. The diagnosis of AKI is mainly based on serum creatinine or urine output, and KDIGO criteria are currently used, but it is known that serum creatinine is a very insensitive indicator,so in the past 20 years, scholars have been exploring biological markers that are more sensitive than blood creatinine and urine output. Humanin is a mitochondrial polypeptide containing 24 amino acids. It was first identified in Alzheimer's disease patients in 2001. Studies have shown that Humanin has a strong mitochondrial protective effect in neurodegenerative diseases, cardiovascular diseases, diabetes, male infertility, cancer and other diseases, and its mechanism may be related to anti-apoptosis, anti-inflammation, regulation of autophagy and maintenance of mitochondrial homeostasis, because Humanin can function through autocrine, paracrine or endocrine forms, so it can be detected in the blood. Studies have shown that Humanin expression in serum or plasma of patients with diabetes and coronary heart disease is declined. Our previous study found the concentration of Humanin in AKI patients was significantly higher than in the normal population.

The goal of this observational study is to explore the value of Humanin for early diagnosis and short-term prognosis of AKI patients after heart transplantation.. The main questions it aims to answer are:whether Humanin can be a novel marker for predicting AKI after heart transplantation

ELIGIBILITY:
Inclusion Criteria:

Guangdong Provincial People's Hospital performs heart transplantation；Adult patients ≥ 18 years of age, male or female；Basic renal function is normal before surgery；The patient's baseline medical records are complete, including basic heart diseases, comorbidities, hemoglobin, renal function, urine protein quantification, serum albumin, lactic acid, C-reactive protein, heart transplantation operation time, preoperative and postoperative medication and blood pressure, blood transfusion history, ICU length of stay, cardiac ultrasound (including LVEF), etc；

Exclusion Criteria:

Age< 18 years；Baseline data were missing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart transplant patients from Guangdong Provincial People's Hospital from September 2022 to May 2024
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Humanin concentration | 3 months
  Highest measured value used
Serum creatinine concentration | 3 months
  Meets KDIGO's definition of AKI

CONTACTS AND LOCATIONS:
Overall Officials: zhilian PP li, doctor, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangdong, Guangzhou, China

DOCUMENTS (1):
  • Study Protocol (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT06125249/Prot_000.pdf